CLINICAL TRIAL: NCT07023757
Title: Effect of Age on PRF Quality; Assessed by Evaluating Healing Outcomes of ARP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Muhammad Saleh, Clinical Assistant Professor, Periodontics and Oral Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00264197
Record Dates: First submitted 2025-06-04; First posted 2025-06-17 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Healing Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet-rich fibrin group. (Active Comparator): Following extraction, a Platelet-rich fibrin plug will be placed in the extraction socket and covered with a collagen plug.
  Interventions: Procedure: Socket preservation
- Collagen plug only (Sham Comparator): Collagen plug only
  Interventions: Procedure: Socket preservation

INTERVENTIONS:
Procedure: Socket preservation — After tooth extraction, the extraction socket will be filled with a collagen plug in one group or a platelet-rich fibrin plug in the other.

SUMMARY:
This study will examine whether using PRF and your age are going to affect the healing and regeneration benefits gained from PRF.

DETAILED DESCRIPTION:
Platelet-rich fibrin (PRF) is commonly used to enhance gum tissue healing and reducing pain after tooth extraction and before placing a dental implant. 44 patients requiring a tooth extraction will be recruited and randomized to receive a collagen plug with or without platelet-rich fibrin.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 20 to 80 years.
2. Patients must require tooth extraction (molars) as a result of caries, periodontal disease, tooth fracture or deemed unrestorable.
3. Non-infected sockets with intact buccal bone (≥1.5 mm in thickness measured through calipers)
4. Patients interested in implant placement following tooth extraction.

Exclusion Criteria:

1. Allergies or hypersensitivities to study related medications.
2. Hematologic disorders/blood dyscrasias.
3. Active infectious diseases of any kind.
4. Liver or kidney dysfunction/failure.
5. Uncontrolled diabetes (HbA1c > 8).
6. Active cancer treatment - such as active chemotherapy or radiation therapy.
7. Taking medications that will affect their bone healing (for example, bisphosphonates, Long-term NSAIDs use, Steroid).
8. Metabolic bone diseases that affect bone healing such as osteoporosis.
9. Pregnant or lactating women (self-reported).
10. Smoke 10 or more cigarettes per day (self-reported).
11. Poor oral hygiene.
12. Systemic diseases that compromise the immune system
13. Anti-coagulant therapy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Alveolar ridge dimension changes | 4 months
  Digitally measured alveolar ridge dimension changes in mm^2 using cone-beam computed tomography
Soft tissue dimension changes | 4 months
  Digitally measured soft tissue changes in mm^2 using intraoral scans

SECONDARY OUTCOMES:
Histological bone density. | 4 months
  Histomorphometry.
Presence of bone turnover proteins. | 4 months
  Immunohistochemistry.
Amount of growth factors | At baseline surgery
  Growth factors (PDGF, VEGF and TGF b1) from PRF obtained from drawn blood
Wound healing index | 1 week, 2 weeks, 4 weeks, and 8 weeks
  Wound healing index (WHI) according to the following scheme: Score "1" for uneventful wound healing with no gingival edema, erythema, suppuration, discomfort or barrier exposure; Score "2" for uneventful wound healing with slight gingival edema, erythema, or discomfort but no suppuration; Score "3" for poor wound healing with significant gingival edema, erythema, discomfort, loss of barrier or any suppuration.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Saleh, BDS, MSD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No